CLINICAL TRIAL: NCT03026166
Title: A Phase 1/2 Study on the Safety of Rovalpituzumab Tesirine Administered in Combination With Nivolumab or Nivolumab and Ipilimumab for Adults With Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study of Rovalpituzumab Tesirine Administered in Combination With Nivolumab and With or Without Ipilimumab for Adults With Extensive-Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment was stopped after the dose-limiting toxicity (DLT) evaluation phase of Cohort 2.
Sponsor: AbbVie (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M16-300; 2016-003686-26 (EudraCT Number)
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Small Cell Lung Cancer
Keywords: Cancer; Extensive-Stage Small Cell Lung Cancer; Nivolumab; Ipilimumab; Rovalpituzumab tesirine
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms | interventions — Ipilimumab; Nivolumab; rovalpituzumab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rovalpituzumab Tesirine and Nivolumab (Experimental): Participants will receive 2 doses of 0.3 mg/kg rovalpituzumab tesirine by intravenous (IV) infusion 6 weeks apart (Day 1 of Cycles 1 and 3), and 2 doses of 360 mg nivolumab IV 3 weeks apart beginning on Cycle 2 (Day 1 of Cycles 2 and 3).
  Participants will then receive maintenance therapy with 480 mg nivolumab IV once every 4 weeks from Cycle 4 until disease progression.
  Interventions: Drug: Nivolumab; Drug: Rovalpituzumab tesirine
- Rovalpituzumab Tesirine and Nivolumab + Ipilimumab 1 mg/kg (Experimental): Participants will receive 2 doses of 0.3 mg/kg rovalpituzumab tesirine IV 6 weeks apart (Day 1 of Cycles 1 and 3), nivolumab 1 mg/kg every 3 weeks for 4 cycles beginning on Cycle 2 (Day 1 of Cycles 2-5), and ipilimumab 1 mg/kg IV every 3 weeks for 4 cycles beginning on Cycle 2 (Day 1 of Cycles 2-5).
  After a 6-week washout, participants will then receive maintenance therapy with 480 mg nivolumab IV once every 4 weeks from Cycle 6 until disease progression.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Rovalpituzumab tesirine
- Rovalpituzumab Tesirine and Nivolumab + Ipilimumab 3 mg/kg (Experimental): Participants will receive 2 doses of 0.3 mg/kg rovalpituzumab tesirine IV 6 weeks apart (Day 1 of Cycles 1 and 3), nivolumab 1 mg/kg every 3 weeks for 4 cycles beginning on Cycle 2 (Day 1 of Cycles 2-5), and ipilimumab 3 mg/kg IV every 3 weeks for 4 cycles beginning on Cycle 2 (Day 1 of Cycles 2-5).
  After an 8-week washout, participants will then receive maintenance therapy with 480 mg nivolumab IV once every 4 weeks from Cycle 6 until disease progression.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Rovalpituzumab tesirine

INTERVENTIONS:
Drug: Ipilimumab — Administered by intravenous infusion
  Other Names: Yervoy®
  Arms: Rovalpituzumab Tesirine and Nivolumab + Ipilimumab 1 mg/kg; Rovalpituzumab Tesirine and Nivolumab + Ipilimumab 3 mg/kg
Drug: Nivolumab — Administered by intravenous infusion
  Other Names: Opdivo®
Drug: Rovalpituzumab tesirine — Administered by intravenous infusion
  Other Names: SC16LD6.5

SUMMARY:
The purpose of this study is to assess the safety and efficacy of rovalpituzumab tesirine administered in combination with nivolumab or nivolumab and ipilimumab in participants with extensive-stage small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
The study planned to enroll three cohorts with approximately 30 participants in each, including a dose-limiting toxicity (DLT) evaluation phase (the first 12 weeks of any treatment) and an expansion phase. Initially, up to 12 participants were to be enrolled into Cohort 1 in order to obtain 6 evaluable participants through the DLT evaluation period of 12 weeks. Safety data were reviewed by a Safety Monitoring Committee (SMC) for each cohort during the DLT evaluation phase before the next cohort opened. Once a new cohort was opened, the previously opened cohort was permitted to continue enrolling participants for the expansion phase for a total of 30 participants per cohort.

Only two of the planned three cohorts enrolled participants in the study based on the SMC recommendation after DLTs were identified in Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically confirmed extensive-stage small cell lung cancer (SCLC) with progressive disease after at least one platinum-based chemotherapeutic regimen and with evaluable or measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* Has active, known, or suspected autoimmune disease
* Had prior exposure to an immuno-oncology or pyrrolobenzodiazepine (PBD)-based drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (35):
- United States (15):
  - Ucsd /Id# 161030, La Jolla, California
  - Florida Hospital /ID# 161017, Orlando, Florida
  - University Cancer & Blood Cent /ID# 161028, Athens, Georgia
  - University of Chicago /ID# 161006, Chicago, Illinois
  - The University of Kansas Clini /ID# 162915, Fairway, Kansas
  - Washington University-School of Medicine /ID# 161011, St Louis, Missouri
  - Rutgers Cancer Institute of NJ /ID# 161032, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center /ID# 161010, New York, New York
  - Duke University Medical Center /ID# 161009, Durham, North Carolina
  - Oregon Health and Science University /ID# 161029, Portland, Oregon
  - Medical University of South Carolina /ID# 161007, Charleston, South Carolina
  - Tennessee Oncology, PLLC /ID# 161012, Nashville, Tennessee
  - Vanderbilt University Med Ctr /ID# 162916, Nashville, Tennessee
  - Virginia Cancer Institute /ID# 161025, Richmond, Virginia
  - University of Wisconsin Clinic /ID# 161013, Madison, Wisconsin
- France (6):
  - CHU de Besancon - Jean Minjoz /ID# 165173, Besançon, Doubs
  - Centre Oscar Lambret /ID# 165169, Lille, Hauts-de-France
  - Institut Gustave Roussy /ID# 165168, Villejuif, Val-de-Marne
  - Institut Sainte Catherine /ID# 165172, Avignon
  - CHRU de Brest - Hospital Morva /ID# 165170, Brest
  - Hopital La Timone /ID# 165171, Marseille
- Germany (4):
  - KH Martha-Maria Halle Dolau /ID# 165180, Halle, Saxony-Anhalt
  - Asklepios Fachkliniken M. Gaut /ID# 165183, Gauting
  - Lungen Clinic Grosshansdorf /ID# 165182, Großhansdorf
  - Lungenfachklinik Immenhausen /ID# 165181, Immenhausen
- Italy (5):
  - Istituto Clinico Humanitas /ID# 165176, Rozzano, Milano
  - Centro di Riferimento Oncologi /ID# 165174, Aviano
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele /ID# 165178, Catania
  - Istituto Europeo di Oncologia /ID# 165175, Milan
  - AO Univ di Modena /ID# 165177, Modena
- Spain (5):
  - Clinica Universitar de Navarra - Pamplona /ID# 165165, Pamplona, Navarra, Comunidad
  - Hosp Univ Quiron Dexues /ID# 165166, Barcelona
  - Hospital Genl Gregorio Maranon /ID# 165162, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 165164, Madrid
  - Hospital Universitario Madrid /ID# 165163, Madrid

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 17 clinical study sites in 4 countries: United States, France, Italy, and Germany.
Pre-assignment Details: Three study cohorts were planned to enroll approximately 30 participants in each, including a dose-limiting toxicity (DLT) evaluation phase (the first 12 weeks of any treatment for all participants) and an expansion phase. However, Cohort 2 was limited to 12 participants and Cohort 3 was not opened.
Groups:
- Rovalpituzumab Tesirine and Nivolumab: Participants received 2 doses of 0.3 mg/kg rovalpituzumab tesirine by intravenous (IV) infusion 6 weeks apart (Day 1 of Cycles 1 and 3), and 2 doses of 360 mg nivolumab IV 3 weeks apart beginning on Cycle 2 (Day 1 of Cycles 2 and 3).
  Participants then received maintenance therapy with 480 mg nivolumab IV once every 4 weeks from Cycle 4 until disease progression.
- Rovalpituzumab Tesirine and Nivolumab + Ipilimumab: Participants received 2 doses of 0.3 mg/kg rovalpituzumab tesirine IV 6 weeks apart (Day 1 of Cycles 1 and 3), nivolumab 1 mg/kg every 3 weeks for 4 cycles beginning on Cycle 2 (Day 1 of Cycles 2-5), and ipilimumab 1 mg/kg IV every 3 weeks for 4 cycles beginning on Cycle 2 (Day 1 of Cycles 2-5).
  After a 6-week washout, participants then received maintenance therapy with 480 mg nivolumab IV once every 4 weeks from Cycle 6 until disease progression.
Period: Overall Study
Arm/Group | Rovalpituzumab Tesirine and Nivolumab | Rovalpituzumab Tesirine and Nivolumab + Ipilimumab
Started | 30 | 12
Completed | 0 | 0
Not Completed | 30 | 12
Not completed — Death | 22 | 7
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Study Terminated by Sponsor | 3 | 3
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rovalpituzumab Tesirine and Nivolumab | Rovalpituzumab Tesirine and Nivolumab + Ipilimumab | Total
Number analyzed (Participants) | 30 | 12 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.87 (8.195) | 57.25 (14.085) | 60.55 (10.256)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 0 | 1 | 1
  ≥ 40 to < 60 years | 11 | 5 | 16
  ≥ 60 years | 19 | 6 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 16 | 7 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 28 | 11 | 39
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29 | 10 | 39
  Black or African American | 1 | 1 | 2
  Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT)
Description: Dose-limiting toxicities were defined as any of the following in the 12-week DLT-evaluation period, graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03:
  * Grade 4 thrombocytopenia (or Grade 3 thrombocytopenia with bleeding) lasting more than 7 days and/or requiring platelet transfusion
  * Grade 4 neutropenia lasting more than 7 days, and/or requiring hematopoietic growth factor rescue, or any febrile neutropenia (Grade 3 or 4 neutropenia with concurrent fever ≥ 38.3°C)
  * Grade 4 anemia unrelated to underlying disease
  * Clinically significant Grade 3 or 4 non-hematologic laboratory abnormality that did not resolve to Grade 0/1 or baseline within 7 days
  * Grade 3 or 4 non-laboratory adverse event (AE), except fatigue, asthenia, nausea, or other manageable constitutional symptom
Time Frame: Up to 12 weeks
Population: DLT-evaluable participants were those who completed 4 cycles treatment during the DLT period or stopped treatment earlier due to DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Rovalpituzumab Tesirine and Nivolumab | Rovalpituzumab Tesirine and Nivolumab + Ipilimumab
Number analyzed (Participants) | 6 | 6
Participants | 1 | 3

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: The investigator rated the severity of each AE according to the NCI CTCAE Version 4.03 and according to the following:
  Grade 1: The AE is transient and easily tolerated by the subject (mild).
  Grade 2: The AE causes the subject discomfort and interrupts the subject's usual activities (moderate).
  Grade 3/4: The AE causes considerable interference with the subject's usual activities and may be incapacitating or life-threatening (severe).
  Grade 5: The AE resulted in death of the subject (severe).
  The maximum severity AE for each participant is reported.
  A serious adverse event was defined as an AE meeting any of the following:
  * Death
  * Life-threatening
  * Resulted in hospitalization or prolongation of hospitalization
  * Resulted in congenital abnormality
  * Resulted in persistent or significant disability or incapacity
  * Was an important medical event requiring medical intervention to prevent a serious outcome.
  Relationship to study drug was assessed by the Investigator.
Time Frame: From the first dose of study drug until 100 days after the last dose of study drug; median duration of treatment was 65 days and 53 days in each cohort respectively.
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rovalpituzumab Tesirine and Nivolumab | Rovalpituzumab Tesirine and Nivolumab + Ipilimumab
Number analyzed (Participants) | 30 | 12
Participants
  Any adverse event | 30 | 12
  Drug-related adverse event | 29 | 12
  Serious adverse event | 23 | 9
  Drug-related serious adverse event | 13 | 6
  Grade 3 adverse event | 11 | 7
  Grade 4 adverse event | 1 | 1
  Grade 5 adverse event | 14 | 4
  Drug-related Grade 3 adverse event | 9 | 10
  Drug-related Grade 4 adverse event | 3 | 1
  Drug-related Grade 5 adverse event | 4 | 0
  AE leading to study drug withdrawal | 12 | 6
  AE leading to treatment interruption | 18 | 8
  AE leading to dose reduction | 0 | 1
  Drug-related AE leading to study drug withdrawal | 9 | 4
  Drug-related AE leading to treatment interruption | 17 | 8
  Drug-related AE leading to dose reduction | 0 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Treatment response was assessed by radiographic tumor evaluations conducted by a central radiology review.
  Objective response rate (ORR) is defined as the percentage of participants whose best overall response is either a confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria for Solid Tumors (RECIST) v1.1.
  Complete response (CR): Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm.
  Partial response (PR): A ≥ 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  CR or PR must have been confirmed at least 4 weeks (28 days) from the initial determination per RECIST v 1.1.
Time Frame: Cohort 1: at Week 6, Week 13, and every 8 weeks thereafter; Cohort 2: at Week 6, Week 12, Week 18, and every 8 weeks thereafter, to the end of follow-up; median duration on follow-up was 31.7 and 48.0 weeks in each cohort respectively.
Population: The Efficacy Analysis Set includes participants who received at least one dose of study drug, had a target lesion identified at Baseline, and either had at least 1 post-dose tumor assessment or discontinued treatment due to AE, progressive disease (PD) or death.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rovalpituzumab Tesirine and Nivolumab | Rovalpituzumab Tesirine and Nivolumab + Ipilimumab
Number analyzed (Participants) | 29 | 11
percentage of participants | 27.6 [12.7 to 47.2] | 36.4 [10.9 to 69.2]

4. Secondary Outcome: Duration of Response (DOR)
Description: Duration of overall response is defined as the time from the date of first documented CR or PR, assessed by central radiology review and based on RECIST v. 1.1, to the documented date of progressive disease (PD) or death, whichever occurred first. Participants who neither progressed nor died were censored at the last evaluable disease assessment. Duration of response was evaluated using Kaplan-Meier methodology.
  Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, with an absolute increase of at least 0.5 cm, or the unequivocal progression of non-target lesions, or the appearance of one or more new lesions.
Time Frame: Cohort 1: at Week 6, Week 13, and every 8 weeks thereafter; Cohort 2: at Week 6, Week 12, Week 18 and every 8 weeks thereafter, to the end of follow-up; median duration on follow-up was 31.7 and 48.0 weeks in each cohort respectively.
Population: The analysis includes participants in the Efficacy Analysis Set with a best overall response of unconfirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rovalpituzumab Tesirine and Nivolumab | Rovalpituzumab Tesirine and Nivolumab + Ipilimumab
Number analyzed (Participants) | 10 | 6
months | 3.8 [1.6 to 5.6] | 3.3 [1.4 to NA] — Could not be estimated due to the low number of events

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from the first dose date to the documented date of PD or death, whichever occurred first, based on central radiology review according to RECIST v 1.1. Progression-free survival was evaluated using Kaplan-Meier methodology. Participants who neither progressed nor died were censored at the last evaluable disease assessment.
  Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, with an absolute increase of at least 0.5 cm, or the unequivocal progression of non-target lesions, or the appearance of one or more new lesions.
Time Frame: From first dose of study drug to the end of follow-up; median duration on follow-up was 31.7 and 48.0 weeks in each cohort respectively.
Population: Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rovalpituzumab Tesirine and Nivolumab | Rovalpituzumab Tesirine and Nivolumab + Ipilimumab
Number analyzed (Participants) | 29 | 11
months | 4.8 [3.2 to 5.3] | 4.1 [1.3 to 6.0]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the first dose date to death for any reason. Participants who were still alive were censored at the last known alive date. Overall survival was evaluated using Kaplan-Meier methodology.
Time Frame: as for outcome 5
Population: The Full Analysis Set includes participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rovalpituzumab Tesirine and Nivolumab | Rovalpituzumab Tesirine and Nivolumab + Ipilimumab
Number analyzed (Participants) | 30 | 12
months | 7.4 [5.0 to 9.1] | 11.0 [2.3 to 17.0]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 100 days after the last dose of study drug; median duration of treatment was 65 days and 53 days in each cohort respectively. All-cause mortality is reported through the end of follow-up; maximum time on study was 115 weeks.
Groups:
- Cohort 1: Rovalpituzumab Tesirine and Nivolumab: Participants received 2 doses of 0.3 mg/kg rovalpituzumab tesirine by intravenous (IV) infusion 6 weeks apart (Day 1 of Cycles 1 and 3), and 2 doses of 360 mg nivolumab IV 3 weeks apart beginning on Cycle 2 (Day 1 of Cycles 2 and 3).
  Participants then received maintenance therapy with 480 mg nivolumab IV once every 4 weeks from Cycle 4 until disease progression.
- Cohort 2: Rovalpituzumab Tesirine and Nivolumab + Ipilimumab: Participants received 2 doses of 0.3 mg/kg rovalpituzumab tesirine IV 6 weeks apart (Day 1 of Cycles 1 and 3), nivolumab 1 mg/kg every 3 weeks for 4 cycles beginning on Cycle 2 (Day 1 of Cycles 2-5), and ipilimumab 1 mg/kg IV every 3 weeks for 4 cycles beginning on Cycle 2 (Day 1 of Cycles 2-5).
  After a 6-week washout, participants then received maintenance therapy with 480 mg nivolumab IV once every 4 weeks from Cycle 6 until disease progression.
Arm/Group | Cohort 1: Rovalpituzumab Tesirine and Nivolumab | Cohort 2: Rovalpituzumab Tesirine and Nivolumab + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 26/30 | 8/12
Serious Adverse Events (participants affected / at risk) | 23/30 | 9/12
Other Adverse Events (participants affected / at risk) | 30/30 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Rovalpituzumab Tesirine and Nivolumab (N=30) | Cohort 2: Rovalpituzumab Tesirine and Nivolumab + Ipilimumab (N=12)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Generalised oedema (General disorders) | 1 (2) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Rovalpituzumab Tesirine and Nivolumab (N=30) | Cohort 2: Rovalpituzumab Tesirine and Nivolumab + Ipilimumab (N=12)
Anaemia (Blood and lymphatic system disorders) | 10 (17) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (14) | 5 (7)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 7 (8) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (2)
Hyperthyroidism (Endocrine disorders) | 1 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 2 (2) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Xerophthalmia (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (4)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (9) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (10) | 3 (3)
Asthenia (General disorders) | 5 (14) | 3 (5)
Chest pain (General disorders) | 1 (1) | 2 (2)
Face oedema (General disorders) | 6 (8) | 2 (2)
Fatigue (General disorders) | 11 (14) | 4 (5)
Localised oedema (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 12 (18) | 3 (4)
Pain (General disorders) | 3 (4) | 0 (0)
Pyrexia (General disorders) | 5 (7) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 2 (2)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (5) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (6) | 0 (0)
Amylase increased (Investigations) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (5) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (4) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 9 (11) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipasaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (10) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 4 (6) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (17) | 5 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (13) | 5 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 6 (8) | 2 (2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 7 (10) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (6)
Subacute cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 4 (5) | 0 (0)
Hypotension (Vascular disorders) | 4 (5) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03026166/Prot_SAP_001.pdf